CLINICAL TRIAL: NCT05679479
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled, Loaded Phase III Study on the Safety and Efficacy of Meplazumab for Injection in Severe Patients With COVID-19
Brief Title: Study on the Safety and Efficacy of Meplazumab for Injection in Severe Patients With COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Pacific Meinuoke Bio Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MPZ-III-01-CN
Record Dates: First submitted 2023-01-10; First posted 2023-01-11 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — meplazumab; Injections; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meplzaumb (Experimental): First dose: 0.2 mg/kg - Day 1; second dose: 0.2 mg/kg - Day 8
  Interventions: Biological: Meplazumab for injection
- Placebo (Placebo Comparator): First dose: control - Day 1; second dose: control - Day 8
  Interventions: Other: Normal saline

INTERVENTIONS:
Biological: Meplazumab for injection — Meplazumab is a humanized anti-CD147 immunoglobulin 2 (IgG2) monoclonal antibody which is expected to block the binding of the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) spike protein to the human host-cell-expressed CD147, thereby blocking entry of SARS-CoV-2 into human tissue. This expectation is based on in vitro functional studies using Vero E6 cells infected with SARS-CoV-2 that demonstrated effective meplazumab mediated virus gene copy number inhibition upwards of 90% as evaluated by quantitative polymerase chain reaction. Meplazumab may also inhibit COVID-19 associated cytokine storm syndrome based on inhibition of the pro inflammatory factor Cyclophilin A host-cell CD147 interaction.
  Arms: Meplzaumb
Other: Normal saline — 0.9% normal saline
  Arms: Placebo

SUMMARY:
This is a multicenter, double-blind, randomized, placebo-controlled, loaded Phase III clinical study. This test is in a new coronavirus infection pneumonia diagnosis and treatment plan of 9 (trial version) "(SoC), on the basis of the standard treatments according to the results of clinical studies have been obtained, using a dose of 0.2 mg/kg, and a placebo. The regimen consisted of a single intravenous infusion of Meplazumab or placebo on day 1 (d0) of the treatment period and d7 after initial administration at a dose of 0.2 mg/kg calculated according to body weight. It is expected that 350 subjects will be randomly assigned to Meplazumab or placebo in a 1:1 ratio. Short-term efficacy evaluation was performed for each subject within 28 days after initial administration to determine the therapeutic efficacy and safety of Meplazumab. Long-term follow-up evaluation was performed within 56 days of initial administration to determine the safety of Meplazumab in each subject.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, male or female;
2. Patients with clinically confirmed 2019-ncov infection (severe) in accordance with the National Health Commission's "Diagnosis and Treatment Protocol for novel coronavirus Infection (Trial version 10)";;
3. Agree to use a highly effective non-pharmacologic contraceptive method within 3 months after signing ICF to the end of the trial;
4. Subjects must be able to understand the study and willing to participate in the study, and sign an informed consent form (if the researcher believes that it is in the interests of the subjects to participate in the study, the informed consent form should be signed by the legal guardian of the subjects and explained in the original medical records and other relevant documents).

Exclusion Criteria:

1. Any physical examination results, laboratory abnormalities and/or any medical history of the subject may, in the investigator's judgment, endanger the subject's safety by participating in the study;
2. Use of an anti-coronavirus treatment such as Paxlovid (nematavir/ritonavir combination package) within 3 half-lives before the first dose or during the study period, About 6.05 h at t1/2), Azvudine tablets (about 9 h at t1/2), and monolavir capsules (about 3.3 h at t1/2) h), ambavirumab/romisivir injection (t1/2 about 45 days /75 days), COVID-19 human immunoglobulin (t1/2 about 3-4 weeks) or recovery plasma (t1/2 about 21 days), deuremidvir hydrobromide tablets (t1/2 about 4.80-6.95 hours), senotevir tablets/ritonavir tablets The combination package (t1/2 about 4.14 h), baritinib (t1/2 about 12.5 h), tocilizumab (t1/2 about 21.5 days), remdesivir (t1/2 about 27 h), lenreterivir (t1/2 about 14.9 h), favelavir (t1/2 about 4.5 h) h), 2-deoxy-D-glucose (t1/2 about 50 min), etc.
3. Critically ill patients with clinically confirmed 2019-ncov infection according to the Diagnosis and Treatment Protocol for 2019 novel Coronavirus Infection (Trial version 10) issued by the National Health Commission of the People's Republic of China;
4. Stage 4 severe chronic kidney disease requiring dialysis (i.e., estimated glomerular filtration rate [eGFR] < 30 mL/min/1.73 m2), an increase in serum creatinine of 44.2 μmol/L within 7 days, oliguria (< 400 mL/24 hours) or anuria (< 100 mL/24 hours);
5. During pregnancy or lactation;
6. They will be transferred to another hospital other than the study site within 72 hours;
7. Known to be allergic to the test drug and its components;
8. No live vaccine (live attenuated vaccine) was administered within 2 weeks before randomization or during study treatment and safety follow-up;
9. Subjects participating in another clinical study at the same time. A washout period of 5 half-lives is required (depending on the study drug or 30 days from any previous study, whichever is longer);
10. Total bilirubin (TBL) > 2× upper limit of normal (ULN), alanine aminotransferase (ALT) > 5×ULN, aspartate aminotransferase (AST) > 5×ULN, or alkaline phosphatase > 5×ULN;
11. Platelet count < 50×109/L or hemoglobin < 70 g/L;
12. Other factors that the investigator deemed inappropriate for trial entry.

Note: researchers should ensure that participants when screening meets all inclusion/exclusion standard. If a subject's status changes (including laboratory results) between screening and initial dosing and if the subject meets one of the exclusion criteria, the subject shall be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2024-01-19 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-04-18 (Actual)

PRIMARY OUTCOMES:
Mortality | Day 28
  All-cause mortality at day 28 (d28)

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of the Air Force Medical University, Xi'an, China

REFERENCES:
- [Derived] Bian H, Chen L, Zhang Z, Wen AD, Zheng ZH, Song LQ, Yao MY, Liu YX, Zhang XJ, Dong HL, Lian JQ, Pan L, Liu Y, Gu X, Zhao H, Wang JW, Wang QY, Zhang K, Jia JF, Xie RH, Luo X, Fu XH, Jia YY, Hou JN, Tan QY, Chen XX, Yang LQ, Lin YL, Wang XX, Zhang L, Zeng QJ, Li WJ, Wang RX, Zhang Y, Sun XX, Wang B, Yang X, Jiang JL, Li L, Wu J, Yang XM, Zhang H, Shi Y, Chen XC, Tang H, Shi HW, Liu SS, Yang Y, Yang TY, Wei D, Chen ZN, Zhu P. Meplazumab, a CD147 antibody, for severe COVID-19: a double-blind, randomized, placebo-controlled, phase 3 clinical trial. Signal Transduct Target Ther. 2025 Apr 14;10(1):119. doi: 10.1038/s41392-025-02208-9. PMID 40222976